CLINICAL TRIAL: NCT00000826
Title: Effect of Fluconazole, Clarithromycin, and Rifabutin on the Pharmacokinetics of Sulfamethoxazole and Dapsone and Their Hydroxylamine Metabolites
Brief Title: Effect of Fluconazole, Clarithromycin, and Rifabutin on the Pharmacokinetics of Sulfamethoxazole-Trimethoprim and Dapsone and Their Hydroxylamine Metabolites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 283; 11259 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Bacterial Infections; Mycoses; HIV Infections
Keywords: Rifabutin; Trimethoprim-Sulfamethoxazole Combination; AIDS-Related Opportunistic Infections; Dapsone; Drug Interactions; Fluconazole; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Clarithromycin; Sulfamethoxazole-Trimethoprim
MeSH Terms: conditions — Bacterial Infections; Mycoses; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Clarithromycin; Rifabutin; Trimethoprim, Sulfamethoxazole Drug Combination; Dapsone; Fluconazole

INTERVENTIONS:
Drug: Clarithromycin
Drug: Rifabutin
Drug: Sulfamethoxazole-Trimethoprim
Drug: Dapsone
Drug: Fluconazole

SUMMARY:
To determine the effects of fluconazole and either rifabutin or clarithromycin, alone and in combination, on the pharmacokinetics of first sulfamethoxazole-trimethoprim and then dapsone in HIV-infected patients.

Although prophylaxis for more than one opportunistic infection is emerging as a common clinical practice in patients with advanced HIV disease, little is known about possible adverse drug interactions. The need exists to define pharmacokinetics and pharmacodynamic adverse interactions of the many combination prophylactic regimens that may be prescribed.

DETAILED DESCRIPTION:
Although prophylaxis for more than one opportunistic infection is emerging as a common clinical practice in patients with advanced HIV disease, little is known about possible adverse drug interactions. The need exists to define pharmacokinetics and pharmacodynamic adverse interactions of the many combination prophylactic regimens that may be prescribed.

In Part A, patients receive sulfamethoxazole-trimethoprim (SMX/TMP) alone for 2 weeks, then in combination with fluconazole, rifabutin, or both drugs, each over 2-week periods in a randomly assigned order. Patients in Part B receive the same regimens except with clarithromycin substituted for rifabutin. In Part C, patients receive dapsone alone for 2 weeks, then in combination with fluconazole, rifabutin, or both drugs in the same manner as in Part A. Part D patients receive the same regimen as those in Part C, except with clarithromycin substituted for rifabutin. Patients are followed every 2 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral therapy provided patient has been on a stable dose for at least 4 weeks prior to study entry.
* Methadone for drug abuse programs provided patient has been on a stable dose for at least 4 weeks prior to the study.

Patients must have:

* HIV infection.
* CD4 count >= 200 cells/mm3.
* No active opportunistic infection.

Prior Medication:

Allowed:

* Antiretroviral therapy.
* Methadone for drug abuse therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Suspicion of gastrointestinal malabsorption problems (at discretion of investigator).
* Known hypersensitivity to dapsone, SMX, or other sulfonamides, trimethoprim, clarithromycin, rifabutin or other rifamycins, fluconazole, or other azoles.
* G-6-PD deficiency or methemoglobinemia (in Part C and D patients only).

Concurrent Medication:

Excluded:

* Cytolytic agents.
* Amiodarone.
* Anesthetics, general.
* Astemizole.
* Azithromycin.
* Barbiturates.
* Carbamazepine.
* Cimetidine.
* Ciprofloxacin.
* Cisapride.
* Clarithromycin (except as required on study).
* Clotrimazole.
* Dexamethasone.
* Disulfiram.
* Erythromycin.
* Fluoroquinolones.
* Fluoxetine.
* Gestodene.
* Hydrochlorothiazide.
* Hypoglycemics, oral.
* Isoniazid.
* Itraconazole.
* Ketoconazole.
* Levomepromazine.
* Loratadine.
* MAO inhibitors.
* Methoxsalen.
* Miconazole.
* Nafcillin.
* Narcotic analgesics.
* Naringenin.
* Nifedipine.
* Norethindrone.
* Pentazocine.
* Phenothiazines.
* Phenytoin.
* Protease inhibitors.
* Quinidine.
* Ranitidine.
* Rifabutin (except as required on study).
* Rifampin.
* Sedative hypnotics.
* Sulfaphenazole.
* Terfenadine.
* Tranquilizers (unless allowed by investigator).
* Tricyclic and tetracyclic antidepressants.
* Troleandomycin.
* Warfarin.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Prior Medication:

Excluded:

* Cytolytic agents within 5 years prior to study entry.
* Rifabutin and/or rifampin within 4 weeks prior to study entry.
* Fluconazoles or other azoles within 4 weeks prior to study entry.
* Glutathione, glutathione precursors, or related prodrugs within 2 weeks prior to study entry.

Excluded within 72 hours prior to study entry:

* Amiodarone.
* Anesthetics, general.
* Astemizole.
* Azithromycin.
* Cimetidine.
* Ciprofloxacin.
* Cisapride.
* Clarithromycin.
* Dexamethasone.
* Disulfiram.
* Erythromycin.
* Fluoroquinolones.
* Fluoxetine.
* Hydrochlorothiazide.
* Hypoglycemics, oral.
* Isoniazid.
* Levomepromazine.
* Loratadine.
* MAO inhibitors.
* Methoxsalen.
* Nafcillin.
* Narcotic analgesics.
* Naringenin.
* Nifedipine.
* Norethindrone.
* Pentazocine.
* Phenothiazines.
* Phenytoin.
* Protease inhibitors.
* Quinidine.
* Ranitidine.
* Sedative hypnotics.
* Sulfaphenazole.
* Terfenadine.
* Tranquilizers (unless allowed by investigator).
* Troleandomycin.
* Warfarin.

Excluded within 4 weeks prior to study entry:

* Barbiturates.
* Carbamazepine.
* Clotrimazole.
* Gestodene.
* Itraconazole.
* Ketoconazole.
* Miconazole.
* Omeprazole.
* Rifabutin.
* Rifampin.
* Tricyclic and tetracyclic antidepressants.

Prior Treatment:

Excluded:

* Blood transfusion within 1 week prior to study entry.
* Radiation therapy within 5 years prior to study entry.

Active drug or alcohol abuse or dependence that would preclude completion of study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Study Completion 1999-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Unadkat J, Study Chair; Trapnell CB, Study Chair
Locations (2):
- United States (2):
  - Ucsf Aids Crs, San Francisco, California
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Cheng B. Preventing opportunistic infections. PI Perspect. 1995 May;(no 16):14-5. PMID 11362422
- [Result] Winter HR, Trapnell CB, Slattery JT, Jacobson M, Greenspan DL, Hooton TM, Unadkat JD. The effect of clarithromycin, fluconazole, and rifabutin on sulfamethoxazole hydroxylamine formation in individuals with human immunodeficiency virus infection (AACTG 283). Clin Pharmacol Ther. 2004 Oct;76(4):313-22. doi: 10.1016/j.clpt.2004.06.002. PMID 15470330